CLINICAL TRIAL: NCT03859648
Title: Outcomes in Adults With Mixed or Conductive Hearing Loss Implanted With the BONEBRIDGE
Brief Title: BONEBRIDGE Bone Conduction Implant in Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment due to COVID-19
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-EL BB
Record Dates: First submitted 2019-02-12; First posted 2019-03-01 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bone Conduction Implant (Experimental): All subjects will be implanted with the bone conduction implant.
  Interventions: Device: BONEBRIDGE

INTERVENTIONS:
Device: BONEBRIDGE — Bone Conduction Implant

SUMMARY:
Approximately thirty subjects with mixed or conductive hearing loss, meeting FDA-cleared candidacy criteria for the BONEBRIDGE, will be implanted and followed for three (3) months post-activation to assess safety and effectiveness of the BONEBRIDGE implant.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older at the time of implantation
* Conductive or mixed hearing loss, defined as:
* Conductive hearing loss with pure-tone average (PTA) for bone conduction thresholds better than or equal to 25 dB at 500, 1000, 2000 and 3000 Hz
* Mixed hearing loss with PTA for bone conduction thresholds better than or equal to 45dB at 500, 1000, 2000, and 3000 Hz
* Air-bone gap greater than or equal to 30 dB at 500, 1000, 2000, and 3000 Hz
* Ability to benefit from amplification as defined by a monosyllabic (CNC) word score of 30% correct or better
* Bilateral BONEBRIDGE can be considered if the difference in PTA for bone conduction thresholds is 10 dB or less between the right and left ears
* Prior experience with acoustic or bone conduction hearing aids, unless candidate is unable to wear amplification for medical reasons
* Able to complete testing materials in English
* CT scan indicating the patient's anatomy is adequate to enable placement of the implant
* Ability to undergo general anesthesia
* Appropriate motivation and expectation levels
* Stated willingness to comply with all study procedures for the duration of the study

Exclusion Criteria:

* Evidence that hearing loss is retrocochlear in origin
* Skin or scalp condition precluding use of external audio processor
* Suspected cognitive impairment or organic brain dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - The Ohio State Wexner Medical Center University, Columbus, Ohio
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badran K, Bunstone D, Arya AK, Suryanarayanan R, Mackinnon N. Patient satisfaction with the bone-anchored hearing aid: a 14-year experience. Otol Neurotol. 2006 Aug;27(5):659-66. doi: 10.1097/01.mao.0000226300.13457.a6. PMID 16868513
- [Background] Riss D, Arnoldner C, Baumgartner WD, Blineder M, Flak S, Bachner A, Gstoettner W, Hamzavi JS. Indication criteria and outcomes with the Bonebridge transcutaneous bone-conduction implant. Laryngoscope. 2014 Dec;124(12):2802-6. doi: 10.1002/lary.24832. Epub 2014 Aug 20. PMID 25142577
- [Background] Schmerber S, Deguine O, Marx M, Van de Heyning P, Sterkers O, Mosnier I, Garin P, Godey B, Vincent C, Venail F, Mondain M, Deveze A, Lavieille JP, Karkas A. Safety and effectiveness of the Bonebridge transcutaneous active direct-drive bone-conduction hearing implant at 1-year device use. Eur Arch Otorhinolaryngol. 2017 Apr;274(4):1835-1851. doi: 10.1007/s00405-016-4228-6. Epub 2016 Jul 30. PMID 27475796
- [Background] Sprinzl GM, Wolf-Magele A. The Bonebridge Bone Conduction Hearing Implant: indication criteria, surgery and a systematic review of the literature. Clin Otolaryngol. 2016 Apr;41(2):131-43. doi: 10.1111/coa.12484. Epub 2016 Feb 4. PMID 26073720
- [Background] Sprinzl G, Lenarz T, Ernst A, Hagen R, Wolf-Magele A, Mojallal H, Todt I, Mlynski R, Wolframm MD. First European multicenter results with a new transcutaneous bone conduction hearing implant system: short-term safety and efficacy. Otol Neurotol. 2013 Aug;34(6):1076-83. doi: 10.1097/MAO.0b013e31828bb541. PMID 23714710
- [Background] Zernotti ME, Sarasty AB. Active Bone Conduction Prosthesis: Bonebridge(TM). Int Arch Otorhinolaryngol. 2015 Oct;19(4):343-8. doi: 10.1055/s-0035-1564329. PMID 26491482

RESULTS

PARTICIPANT FLOW:
Groups:
- BONEBRIDGE: Subjects implanted with the transcutaneous bone conduction implant
Period: Overall Study
Arm/Group | BONEBRIDGE
Started | 8
Completed | 6
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- BONEBRIDGE: All subjects implanted with the transcutaneous bone conduction implant.
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 47 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This information was not collected from any participant.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race and Ethnicity Not Collected Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 5
  United States | 3
Duration of hearing loss [Mean (Full Range); unit: years] | 28.4 [15 to 65]

OUTCOME MEASURES:

1. Primary Outcome: Number and Proportion of Subjects Experiencing Device Related Adverse Events
Description: Adverse events will be collected and reported throughout the duration of the study.
Time Frame: Up to three (3 months) post activation
Population: One subject did not pursue surgery after baseline evaluation. This subject was removed from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 8
Participants | 1

2. Primary Outcome: Percentage Change in AZ Bio Sentence Score in Noise
Description: Percent improvement in AZ Bio sentence in noise scores will be compared from baseline to 3 months post activation.
Time Frame: Baseline and 3 months post activation
Population: One subject was lost to follow up after 1 month, and one subject did not participate in postoperative intervals due to an adverse event. These subjects were removed from this analysis.
Measure: Mean (Full Range); unit: percent improvement
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 6
percent improvement | 42.2 [23 to 95]

3. Secondary Outcome: Percentage Change in CNC Word Score
Description: Percent improvement in CNC word scores will be compared from baseline to 3 months post activation.
Time Frame: Baseline and 3 months post activation
Population: as for outcome 2
Measure: Mean (Full Range); unit: percent improvement
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 6
percent improvement | 38.3 [23 to 70]

4. Secondary Outcome: Number of Subjects With Stable or Better Soundfield Thresholds
Description: The number of subjects with stable or better aided soundfield thresholds at 3 months post activation compared to baseline unaided soundfield thresholds
Time Frame: Baseline and 3 months post activation
Population: One subject was lost to follow up after 1 month, one subject did not participate in postoperative intervals due to an adverse event, and sound field data was missing for one subject. These subjects were removed from this analysis.
Measure: Number; unit: Participants
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Number of Subjects With Better QuickSIN Signal-to-noise-ratio Performance
Description: The number of subjects with similar or better performance on the QuickSIN (Speech In Noise) task in the implanted ear compared to baseline performance
Time Frame: Baseline and 3 months post activation
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 6
Participants | 6

6. Secondary Outcome: Number of Subjects With Stable Unaided Bone Conduction Thresholds
Description: The number of subjects with stable bone conduction thresholds at the device activation interval compared to pre-operative bone conduction thresholds.
Time Frame: Baseline and 2 weeks post surgery
Population: One subject did not participate in postoperative intervals due to an adverse event. These subjects were removed from this analysis.
Measure: Number; unit: Participants
Arm/Group | BONEBRIDGE
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from surgery through 3 months post-activation.
Arm/Group | BONEBRIDGE
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BONEBRIDGE (N=8)
Postoperative infection (Infections and infestations) | 1 (1) — Postoperative infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BONEBRIDGE (N=8)
Scalp sensitivity (Skin and subcutaneous tissue disorders) | 1 (1) — Scalp sensitivity at implant site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03859648/Prot_SAP_000.pdf